CLINICAL TRIAL: NCT04274335
Title: A Randomised Controlled Trial to Assess the Pharmacokinetics and Pharmacodynamics of Intramuscular, Intravenous and Oral Administration of Tranexamic Acid in Women Giving Birth by Caesarean Section
Brief Title: Pharmacokinetics and Pharmacodynamics of Tranexamic Acid in Women Having Caesarean Section Birth [WOMAN-PharmacoTXA]
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Rawalpindi Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-KEP-401
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2022-08

CONDITIONS: Pregnancy, High Risk
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intravenous tranexamic acid (Experimental)
  Interventions: Drug: Tranexamic Acid 100Mg/Ml Inj Vil 10Ml
- Intramuscular tranexamic acid (Experimental)
  Interventions: Drug: Tranexamic Acid Injectable Product
- Oral liquid tranexamic acid (Experimental)
  Interventions: Drug: Tranexamic Acid Oral Solution
- No tranexamic acid (No Intervention)

INTERVENTIONS:
Drug: Tranexamic Acid 100Mg/Ml Inj Vil 10Ml — 1 gram of tranexamic acid to be administered intravenously
  Arms: Intravenous tranexamic acid
Drug: Tranexamic Acid Oral Solution — 4 grams of tranexamic acid given as an oral solution
  Arms: Oral liquid tranexamic acid
Drug: Tranexamic Acid Injectable Product — 1 gram of tranexamic acid given as 2 separate intramuscular injection
  Arms: Intramuscular tranexamic acid

SUMMARY:
Intramuscular injection and oral solution of tranexamic acid (TXA) would increase its use in situations where administration of intravenous drugs is difficult. The investigators aim to assess the population pharmacokinetics (PK) and pharmacodynamics (PD) of intravenous, intramuscular and oral TXA in women undergoing undergoing caesarean section (CS) with at least one known risk factor for postpartum haemorrhage (PPH)

DETAILED DESCRIPTION:
An open label, randomised controlled trial to assess the pharmacokinetics and pharmacodynamics of intramuscular, intravenous and oral solution administration of tranexamic acid in women giving birth by caesarean section. 120 women (30 receiving oral liquid, 30 receiving intramuscular, 30 receiving intravenous and 30 receiving no TXA who have at least 6 evaluable PK samples will be randomised.

ELIGIBILITY:
Inclusion Criteria:

* Women admitted to hospital giving birth by CS
* History of at least one risk factor for PPH
* Adult (≥18 years old)

Exclusion Criteria:

* Women giving birth vaginally
* Women with a known allergy to TXA or its excipients
* Women with current antepartum haemorrhage
* Women known to have received TXA within 48 hours prior to randomisation
* Women with known renal impairment
* Women with any known blood clotting disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women giving birth by caesarean section
Enrollment: 120 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic | 24 hours after randomisation
  Concentration of TXA in Maternal blood over time

SECONDARY OUTCOMES:
Placenta transfer of TXA | at birth of baby
  Concentrations of TXA in placenta cord blood
Placenta transfer of TXA | within 24 hours of birth
  Concentration of neonate TXA
Concentration of D-dimer | up to 24 hours after randomisation
  Maternal blood concentration over time
Maternal blood volume lost | from incision to 2 hours from CS
  total blood loss
frequency of Injection site reaction from IM administration | from randomisation up to 7 days after
  Local reactions at injection site
Number of Adverse events (maternal and neonate) | from randomisation up to 7 days after
  any untoward medical events
Number of women with a clinical diagnosis of PPH | up to 24 hours after giving birth
  total blood loss of >1000 mL or any blood loss sufficient to cause haemodynamic instability or requires treatment

CONTACTS AND LOCATIONS:
Overall Officials: Haleema Shakur-Still, Study Chair — London School of Hygiene and Tropical Medicine; Ian Roberts, Study Chair — London School of Hygiene and Tropical Medicine
Locations (2):
- MCH PIMS, Islamabad, Pakistan
- Women and Newborn Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Totally anonymised dataset used for main analysis will be made freely available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: freely available 1 year after main publication
Access Criteria: Free login to website required for monitoring usage of data
URL: https://freebird.lshtm.ac.uk

REFERENCES:
- [Derived] Shakur-Still H, Roberts I, Grassin-Delyle S, Chaudhri R, Geer A, Arribas M, Lamy E, Mansukhani R, Lubeya MK, Javaid K, Kayani A, Israr N, Mazhar SB, Urien S, Bouazza N, Foissac F, Prowse D, Carrington L, Barrow C, Onandia JG, Balogun E. Alternative routes for tranexamic acid treatment in obstetric bleeding (WOMAN-PharmacoTXA trial): a randomised trial and pharmacological study in caesarean section births. BJOG. 2023 Sep;130(10):1177-1186. doi: 10.1111/1471-0528.17455. Epub 2023 Apr 5. PMID 37019443
- [Derived] Arribas M, Roberts I, Chaudhri R, Geer A, Prowse D, Lubeya MK, Kayani A, Javaid K, Grassin-Delyle S, Shakur-Still H. WOMAN-PharmacoTXA trial: Study protocol for a randomised controlled trial to assess the pharmacokinetics and pharmacodynamics of intramuscular, intravenous and oral administration of tranexamic acid in women giving birth by caesarean section. Wellcome Open Res. 2021 Jun 16;6:157. doi: 10.12688/wellcomeopenres.16884.1. eCollection 2021. PMID 34250266